CLINICAL TRIAL: NCT05844371
Title: Clinical Efficacy and Safety of Adjuvant Immunotherapy (Tirelizumab) Plus Chemotherapy Versus Adjuvant Chemotherapy Alone in Lymph Node Positive Patients With Gastric Cancer After D2 Radical Resection
Brief Title: Efficacy and Safety of Tirelizumab Plus Chemotherapy Versus Chemotherapy Alone in Patients With Lymph Node Positive Gastric Cancer After Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yixing People's Hospital (Other)
Responsible Party: Principal Investigator, Zhou Yan, Chief physician, Yixing People's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YixingPH
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Drug Therapy; Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- study group (Experimental): chemotherapy with oxaliplatin + heroda regimen (oxaliplatin 130mg / m2 D1, heroda tablets 1000mg / m2 bid d1-14, 21d repeated), during which tirelizumab (200mg, q3w) was used. After 6 cycles of chemotherapy, monotherapy with tirelizumab (200 mg, q3w) was maintained until 1 year.
  Interventions: Drug: tirelizumab; Drug: chemotherapy with oxaliplatin + heroda
- Control group (Active Comparator): 6 cycles of oxaliplatin + heroda regimen chemotherapy.
  Interventions: Drug: chemotherapy with oxaliplatin + heroda

INTERVENTIONS:
Drug: tirelizumab — Tirelizumab (200 mg, q3w) was added and maintained until one year, starting with adjuvant chemotherapy after surgery.
  Arms: study group
Drug: chemotherapy with oxaliplatin + heroda — chemotherapy with oxaliplatin + heroda

SUMMARY:
Lymph node positive patients after D2 radical surgery for gastric cancer, who started to be treated at Yixing people's Hospital in April 2021, were selected and enrolled into the study group according to the patients' wishes: immune (tirelizumab) combined with chemotherapy (XELOX regimen) or control group: chemotherapy alone (XELOX regimen). Each enrolled patient signed an informed consent form approved by the ethics committee, signed, and dated. Efficacy and adverse effects were assessed in both groups.

ELIGIBILITY:
Inclusion criteria：(1) With a good bone marrow reserve, e. g. : leukocytes ≥ 4 × 109 / L, neutrophils ≥ 1.5 × 109 / L, platelets ≥ 100 × 109 / L and hemoglobin ≥ 90 g / L.(2) Cardiopulmonary function was unremarkable.(3) There were no abnormalities in liver and kidney function. For example: creatinine ≤ 1.5 × ULN or a calculated serum creatinine clearance ≥ 50 ml / min (calculated according to the Cockcroft Gault formula), albumin ≥ 30 g / L, and total bilirubin ≤ 1.5 × ULN, alanineaminotransferase (ALT) / aspartate aminotransferase (AST) ≤ 2 × ULN.(4) International normalized ratio / activated partial thromboplastin time ≤ 1.5 × ULN.(5) Age older than 18 years, karonfsky performance status (KPS) score ≥ 80, and premedication patients' bone marrow status, liver and kidney function, and cardiopulmonary function had little impact on prognosis.

Exclusion criteria: Had a previous history of immunodeficiency, or had other acquired, congenital immunodeficiency diseases, or a history of organ transplantation; Preexisting thyroid dysfunction and, with medical therapy, thyroid function still cannot be maintained within the normal range; Women who were pregnant or lactating; Those with a history of substance abuse who are unable to abstain or who have a mental disorder.

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
The 1-year DFS rate | 1 year
  within one year from onset

CONTACTS AND LOCATIONS:
Overall Officials: Yan Zhou, Study Director — Yixing People's Hospital
Locations (1):
- Yixing People's Hospital, Yixing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhang T, Song X, Xu L, Ma J, Zhang Y, Gong W, Zhang Y, Zhou X, Wang Z, Wang Y, Shi Y, Bai H, Liu N, Yang X, Cui X, Cao Y, Liu Q, Song J, Li Y, Tang Z, Guo M, Wang L, Li K. The binding of an anti-PD-1 antibody to FcgammaRIota has a profound impact on its biological functions. Cancer Immunol Immunother. 2018 Jul;67(7):1079-1090. doi: 10.1007/s00262-018-2160-x. Epub 2018 Apr 23. PMID 29687231
- [Result] Lee SH, Lee HT, Lim H, Kim Y, Park UB, Heo YS. Crystal structure of PD-1 in complex with an antibody-drug tislelizumab used in tumor immune checkpoint therapy. Biochem Biophys Res Commun. 2020 Jun 18;527(1):226-231. doi: 10.1016/j.bbrc.2020.04.121. Epub 2020 May 1. PMID 32446372
- [Result] Shen L, Guo J, Zhang Q, Pan H, Yuan Y, Bai Y, Liu T, Zhou Q, Zhao J, Shu Y, Huang X, Wang S, Wang J, Zhou A, Ye D, Sun T, Gao Y, Yang S, Wang Z, Li J, Wu YL. Tislelizumab in Chinese patients with advanced solid tumors: an open-label, non-comparative, phase 1/2 study. J Immunother Cancer. 2020 Jun;8(1):e000437. doi: 10.1136/jitc-2019-000437. PMID 32561638
- [Derived] Shi JW, Zhou Y, Wu S. Clinical efficacy and safety of adjuvant immunotherapy (Tislelizumab) plus chemotherapy vs. adjuvant chemotherapy alone in lymph node-positive patients with gastric cancer after D2 radical resection: a prospective, 2-arm, phase II study. Eur Rev Med Pharmacol Sci. 2023 Nov;27(21):10472-10480. doi: 10.26355/eurrev_202311_34324. PMID 37975371